CLINICAL TRIAL: NCT03030443
Title: Patient Preferences in Anesthesia for Abortion Care
Acronym: PAC
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Rameet Singh, Chief, Division of Family Planning, University of New Mexico
Other Study IDs: 16-275
Record Dates: First submitted 2017-01-10; First posted 2017-01-25 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Pregnancy Termination in First Trimester
Keywords: Pain management; Nitrous
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Oral Sedation: Patients in this group will receive a standard procedure first trimester abortion using oral sedation for pain management following the clinic's protocol.
  Patients in both groups will be administered a Visual Analog Scale (VAS) assessing pain on an unmarked 100mm VAS scale with anchors at 0mm (left) being "no pain" and 100mm (right) being "pain as bad as it could be" before their procedure and immediately following procedure completion.
- Nitrous Oxide: Patients in this group will receive a standard procedure first trimester abortion using titrated nitrous oxide for pain management following the clinic's protocol.
  Patients in both groups will be administered a Visual Analog Scale (VAS) assessing pain on an unmarked 100mm VAS scale with anchors at 0mm (left) being "no pain" and 100mm (right) being "pain as bad as it could be" before their procedure and immediately following procedure completion.

SUMMARY:
This study will use semi-structured interviews with participants in a prospective cohort study to explore women's experiences of pain and preferences in pain management during first trimester surgical abortion to create a more patient centered experience. We will analyze two study cohorts of women undergoing first trimester surgical abortion: women choosing oral anesthesia and women choosing nitrous oxide.

DETAILED DESCRIPTION:
This study will utilize an open-ended semi-structured interview format to elicit a broader understanding of the multi-dimensional pain experience of woman undergoing an abortion procedure. This study seeks to provide further evaluation of the pain experience and preferences of women receiving alternative methods of pain management such as oral sedation and nitrous oxide.

The study will use semi-structured interviews to explore women's experiences of pain and preferences in pain management during first trimester surgical abortion and will include a procedural pain outcome using the visual analog scale (VAS) to create a more patient centered experience.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing first trimester surgical abortion choosing between oral anesthesia or nitrous oxide for pain management
* women who are able to read and understand English
* women who are 18 years old or older

Exclusion Criteria:

* under the age of 18
* women unable to consent and/or are cognitively impaired
* women who are incarcerated
* women who do not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women undergoing first trimester surgical abortion choosing between oral anesthesia and nitrous oxide. All patients will be English-speaking women who are 18 years old or older.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-23 (Actual)

PRIMARY OUTCOMES:
Identify Patient Priorities and Preferences for pain and pain management through Qualitative Analysis | through patient completion in study, up to one week following the procedure
  To identify patient priorities and preferences for pain and pain management using Qualitative Analysis prior to their first trimester surgical abortion under local anesthesia with oral or nitrous oxide sedation.

SECONDARY OUTCOMES:
Compare quantitative and qualitative assessment of pain | through patient completion in study, up to one week following the procedure
  Compare the quantitative objective assessment of maximum procedural pain using the visual analog scale (VAS) with the qualitative assessment of pain obtained via semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Rameet Singh, MD, MPH, Principal Investigator — University of New Mexico Health Sciences Center
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No